CLINICAL TRIAL: NCT03841630
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3437943 in Healthy Subjects
Brief Title: A Safety Study of LY3437943 Given as a Single Injection in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17136; J1I-MC-GZBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY3437943 (Experimental): Escalating doses of LY3437943 administered as an injection under the skin in healthy participants
  Interventions: Drug: LY3437943
- Placebo (Placebo Comparator): Matching placebo administered as an injection under the skin in healthy participants
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3437943 — Administered subcutaneously (SC)
  Arms: LY3437943
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This study is being conducted to determine the side effects related to LY3437943 given as a single injection under the skin to healthy participants. Blood tests will be performed to check how much LY3437943 gets into the bloodstream and how long the body takes to get rid of it. Each enrolled participant will receive a single dose of LY3437943 or placebo. The study will last up to approximately 71 days for each participant, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female who cannot get pregnant
* Have a body mass index (BMI) between 19 and 40 kilograms per square meter (kg/m²), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG, heart tracing), blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for ease of blood sampling

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously completed or withdrawn from this study
* Smoke more than the equivalent of 10 cigarettes per day and are unwilling to stop smoking during the inpatient stay in the study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Have been treated with weight loss medications within 3 months of screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through final follow-up at approximately Day 43
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics: Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-inf]) of LY3437943 | Baseline through final follow-up at approximately Day 43
  Pharmacokinetics: AUC(0-inf) of LY3437943
Pharmacokinetics: Maximum Concentration (Cmax) of LY3437943 | Baseline through final follow-up at approximately Day 43
  Pharmacokinetics: Cmax of LY3437943
Pharmacokinetics: Time to Maximum Concentration (Tmax) of LY3437943 | Baseline through final follow-up at approximately Day 43
  Pharmacokinetics: Tmax of LY3437943

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No